CLINICAL TRIAL: NCT03539835
Title: Resistance Training to Improve Fatigue and Physical Function in Postmenopausal Breast Cancer Survivors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Emory University (Other)
Responsible Party: Principal Investigator, Joe Nocera, Assistant Professor, Emory University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: IRB00103558
Record Dates: First submitted 2018-05-16; First posted 2018-05-29 (Actual); Last update posted 2020-07-27 (Actual); Status verified 2020-07

CONDITIONS: Cancer
Keywords: Breast Cancer Survivors; Resistance Training; Fatigue; Physical Function; Behavioral Function; Kynurenine metabolism
MeSH Terms: conditions — Neoplasms; Fatigue | interventions — Resistance Training

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Resistance training (Experimental)
  Interventions: Other: Resistance training (RT)
- Cognitively-based compassion training (Active Comparator)
  Interventions: Behavioral: Cognitively-based compassion training control (CBCT)

INTERVENTIONS:
Other: Resistance training (RT) — Resistance training (RT) will include 15 repetitions for two sets and to exhaustion on the third set for seven major muscle groups: the leg and chest press, knee extension, leg curl, row, abdominal crunch, and bicep curl. Resistance is gradually increased to account for strength gains when subjects are able to complete 20 repetitions on the third set.
  Arms: Resistance training
Behavioral: Cognitively-based compassion training control (CBCT) — Cognitively-based compassion training control (CBCT) classes will be performed in a group setting for 1.5-2 hours per week, and consist of didactics, class discussion, and guided meditation practice. Each class will begin with a period of meditation to calm and focus the mind, followed by analytical practices designed to challenge unexamined assumptions regarding feelings, and actions toward others with a focus on generating spontaneous empathy and compassion for themselves and others.
  Arms: Cognitively-based compassion training

SUMMARY:
This study will begin to fill a knowledge gap by determine whether changes in kynurenine metabolism occur following Resistance Training (RT) and relate to reductions in inflammation and improved behavioral and physical function as this may identify potential targets for interventions to promote cancer recovery.

DETAILED DESCRIPTION:
Interventions that reduce pro-inflammatory cytokines with resultant stimulation of kynurenine metabolism may be increasingly important in Breast Cancer Survivors (BCS) to prevent susceptibility to cancer associated fatigue, depression, and declines in muscle mass and function.

There is emerging evidence that supports exercise as a non-pharmacological therapy to prevent cancer recurrence, sedentary behaviors, and obesity during cancer survivorship . It seems that interventions that include resistance training (RT) are most efficacious at reducing fatigue in BCS This study will begin to fill a knowledge gap by determine whether changes in kynurenine metabolism occur following RT and relate to reductions in inflammation and improved behavioral and physical function as this may identify potential targets for interventions to promote cancer recovery.

ELIGIBILITY:
Inclusion Criteria:

1. within 6 months to 10 years post active breast cancer therapy (i.e. surgery/chemotherapy) for stage I-III invasive breast cancer,
2. at least 6 months post breast reconstruction (if applicable),
3. lack of menses for at least one year,
4. BMI 20-35 kg/m2,
5. fatigued (subjective reporting ≥3 on a 1-10 scale),
6. untrained with regard to structured resistance training (no more than 3x/week).

Exclusion Criteria:

1. plans for surgery (e.g., breast reconstruction) during the study period,
2. taking an anticoagulant medication (i.e. heparin, apixaban, rivaroxaban),
3. allergic to lidocaine,
4. orthopedic or chronic pain condition restricting exercise,
5. Mini-Mental Status Examination (MMSE) scores below education-specific cut-points (less than 23 for more than 9th grade education and less than 17 for less than 8th grade education),
6. unable to receive physician medical clearance.

Ages: 50 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Female
Enrollment: 28 (Actual)
Dates: Start 2018-12-10 (Actual); Primary Completion 2020-03-09 (Actual); Study Completion 2020-03-12 (Actual)

PRIMARY OUTCOMES:
Change in fatigue assessed by Multidimensional Fatigue Inventory (MFI) score | Baseline, 12 weeks follow up
  The Multidimensional Fatigue Inventory (MFI) is a 20-item self-report instrument designed to measure fatigue. It covers the following dimensions: General Fatigue, Physical Fatigue, Mental Fatigue, Reduced Motivation and Reduced Activity. Each scale contains four items for which the person had to indicate on a seven-point scale to what extent the particular statement applies to him or her. An equal number of items is worded in a positive and in a negative direction to counteract response tendencies.

SECONDARY OUTCOMES:
Change in depression assessed by Hamilton Depression Rating Scale (HAM-D) score | Baseline, 12 weeks follow up
  Although the HAM-D form lists 21 items, the scoring is based on the first 17. Eight items are scored on a 5-point scale, ranging from 0 = not present to 4 = severe. Nine are scored from 0-2.
Change in balance test score | Baseline, 12 weeks follow up
  Berg Balance Scale is an observer rated scale developed to rate fall risk that consists of 14 items (0-4 point scale) of mobility related to balance.
Change in muscle function assessed by Isometric Handgrip test. | Baseline, 12 weeks follow up
  Hand grip strength of both arms will be assessed using a handheld dynamometer. The subjects will be tested while seated with the shoulders adducted, the elbow flexed to 90 degrees, and the forearm in a neutral position. The subjects will be instructed to "squeeze as hard as possible" during 3-5 second efforts.
Change in muscle function assessed by Lower Extremity Endurance test | Baseline, 12 weeks follow up
  The subjects will be asked to perform the leg press and leg extension exercises at 60% of maximum strength as many times as they can before fatigue, paced by a metronome set to 30. Endurance in the right and left legs will be tested separately using equipment that is built to isolate single leg movement.
Change in muscle function assessed by Lower Extremity Strength test | Baseline, 12 weeks follow up
  Standardized strength assessment protocol that includes 4-6 trials with rest periods of the leg extension, leg press, and chest press exercises will be used. Strength in the right and left legs will be tested separately.
Change in Timed Up and Go (TUG) completion time | Baseline, 12 weeks follow up
  Subjects are observed and timed while they rise from a chair, walk 3 meters, turn around, walk back, and sit down. The total time to complete this task will be recorded.
Change in 30 meter walk velocity | Baseline, 12 weeks follow up
  Self-selected and fastest-comfortable floor walking velocity will be determined from 30 meter walks with subjects using the same assistive device and/or orthosis as normally used to "walk across the room at home."
Change in Functional Gait Assessment score | Baseline, 12 weeks follow up
  Subjects will be asked to perform various tasks to assess functional gait including stepping onto a small stool, doing a turn, and picking a small object off the floor. Participants will be scored on their ability to perform each task without difficulty. A total score out of a maximum of 30 points will be reported.
Change in 6 min walk distance | Baseline, 12 weeks follow up
  Subjects will use the same assistive device typically used and will be instructed to cover as much distance as they can in six minutes over a flat walking surface.
Change in Resting Metabolic Rate (RMR) | Baseline, 12 weeks follow up
  RMR will be measured using the ventilated hood technique while subjects lie quietly in bed for 30-45 mins under a clear plastic hood with expired air collected through a one-way valve. RMR will be measured at rest under fasting conditions. It will be reported as a continuous variable of kilocalories/day.
Change in peroxisome proliferator-activated receptor gamma coactivator 1-alpha (PGC-1α) level | Baseline, 12 weeks follow up
  Peroxisome proliferator-activated receptor gamma coactivator 1-alpha (PGC-1α) is a key transcription coactivator regulating energy metabolism in a tissue-specific manner. PGC-1α level will be measured by enzyme-linked immunosorbent assay in blood sample.
Change in kynurenic acid level | Baseline, 12 weeks follow up
  Kynurenic acid is a product of the normal metabolism of amino acid L-tryptophan. It has been shown that kynurenic acid possesses neuroactive activity. Kynurenic acid level will be measured by enzyme-linked immunosorbent assay in blood sample. .
Change in interleukin-6 (IL-6) level | Baseline, 12 weeks follow up
  IL-6 is an interleukin that acts as both a pro-inflammatory cytokine and an anti-inflammatory marker in skeletal muscle. IL-6 level will be measured by enzyme-linked immunosorbent assay in blood sample.
Change in tumor necrosis factor-α (TNF-α) protein level | Baseline, 12 weeks follow up
  tumor necrosis factor-α (TNF-α) is a cell signaling protein (cytokine) involved in systemic inflammation and is one of the cytokines that make up the acute phase reaction.TNF-α protein level will be measured by enzyme-linked immunosorbent assay in blood sample.

CONTACTS AND LOCATIONS:
Overall Officials: Monica Serra, MD, Principal Investigator — Emory University
Locations (1):
- Winship Cancer Institute, Atlanta, Georgia, United States

IPD SHARING:
Plan to Share IPD: No